CLINICAL TRIAL: NCT00732186
Title: Phase Ib Study Evaluating the Safety and Exploring the Molecular and Cytogenetic Response of Combination Therapy With Dasatinib and Ipilimumab in Patients With Chronic or Accelerated Phase Chronic Myeloid Leukemia
Brief Title: Study of Ipilimumab and Dasatinib Combination Therapy in Patients With Chronic or Accelerated Chronic Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA184-033
Record Dates: First submitted 2008-08-07; First posted 2008-08-11 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2009-11

CONDITIONS: Leukemia, Myeloid, Chronic
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Group 1 and Group 2 (Experimental)
  Interventions: Biological: Ipilimumab

INTERVENTIONS:
Biological: Ipilimumab — IV Solution, IV, 10 mg/kg, (if dose reduction necessary at 3 mg/kg), Every three weeks for the first 10 weeks, with a booster at week 22, Up to 38 weeks depending on response
  Other Names: BMS-734016; MDX-010

SUMMARY:
The purpose of the study is to assess the safety of ipilimumab and dasatinib combination therapy in patients with CML

ELIGIBILITY:
Inclusion Criteria:

* Ph+ CML on dasatinib therapy
* Loss of cytogenetic or molecular response while on dasatinib therapy
* On stable dose of dasatinib for a minimum of 12 weeks and with < 14 day interruption of treatment

Exclusion Criteria:

* Blast crisis CML
* Autoimmune disease
* Uncontrolled or significant cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety of ipilimumab in combination with dasatinib in CML patients with a loss of previously achieved major molecular response or a loss of previously achieved cytogenetic response to dasatinib | At weeks 1, 4, 7, 10, 14, 18, 22, 26, 30, 34 and 38

SECONDARY OUTCOMES:
To evaluate the frequency of molecular response, complete cytogenetic response and an overall efficacy signal response rate | At weeks 1, 4, 7, 10, 14, 18, 22, 26, 30, 34 and 38
To explore the immunologic responses to combination therapy with ipilimumab and dasatinib | At weeks 1, 4, 7, 10, 14, 18, 22, 26, 30, 34 and 38
To explore whether molecular responses to combination therapy with ipilimumab and dasatinib correlate with immunologic responses | At weeks 1, 4, 7, 10, 14, 18, 22, 26, 30, 34 and 38

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- The University Of Texas, M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx